CLINICAL TRIAL: NCT02297646
Title: The Influence of Carbohydrates on Training Efficacy and Health Status in Healthy Adults
Brief Title: Influencing Factors on Training Efficacy in Healthy Adults
Acronym: CHO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Anne Krieg M.D., M.D., Universität des Saarlandes
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Saarland University - CHO
Record Dates: First submitted 2013-09-10; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Health Status; Maximal and Submaximal Parameters of Physical Performance
Keywords: Prevention; Exercise; Health; Endurance
MeSH Terms: conditions — Motor Activity | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrates (Experimental): 50 grams of carbohydrates 4 times a week for each training session
  Interventions: Behavioral: Endurance Training
- Control (Placebo Comparator): no carbohydrate intake
  Interventions: Behavioral: Endurance Training

INTERVENTIONS:
Behavioral: Endurance Training
  Other Names: 4 sessions a week at 70 percent heart rate reserve

SUMMARY:
The purpose of this study is to investigate the effects of carbohydrate intake on training efficacy and health parameters of an endurance training program in healthy adults.

DETAILED DESCRIPTION:
Carbohydrate availability in endurance exercise seems to attenuate exercise-induced perturbations of cellular homeostasis and consequently diminishes the stimulus for training adaptation. Therefore, a negative relationship with exercise efficacy seems plausible. However, experimental evidence is rare and far from conclusive. Therefore, the present study aims to test the influence of carbohydrate intake on the efficacy of a typical preventive training program.

ELIGIBILITY:
Inclusion Criteria:

* no diseases
* nonsmoker
* BMI 25-30 kg/m²
* blood pressure <160/100 mm/Hg
* unmedicated
* untrained status
* V̇O2max < 50 mL/kg/min

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum oxygen consumption (VO2max) | 24 weeks
  VO2max

SECONDARY OUTCOMES:
Numerous serum parameters from venous blood (LDL, HDL, Cholesterol, Triglycerides) | 24 weeks
  cardiovascular parameters:
  * LDL
  * HDL
  * Cholesterol
  * Triglycerides
Resting heart rate | 24 weeks
Resting blood pressure | 24 weeks
Body fat (Skinfold thickness) | 24 weeks
  Skinfold thickness
Ventilatory anaerobic threshold (VT) | 24 weeks
  VT

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, M.D. Prof., Principal Investigator — Universität des Saarlandes
Locations (1):
- Institute of Sports and Preventive Medicine, Saarland University, Saarbrücken, Saarland, Germany